CLINICAL TRIAL: NCT06089291
Title: Persona IQ Cohort Study: A Multicentric Prospective Cohort Study of the Persona IQ® Personalized Knee System With the Mymobility® Care Management Application
Brief Title: Persona IQ Cohort Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CLU2021-46TDS
Record Dates: First submitted 2023-09-26; First posted 2023-10-18 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Osteo Arthritis Knee; Knee Arthritis; Monitoring Orthopedic Devices; Total Knee Arthroplasty; Total Knee Replacement
Keywords: Cemented Primary Total Knee Arthroplasty; Medical Device; Performance; Safety; Persona IQ; Remote Therapeutic Monitoring; RTM; CTE; CSE; Smart Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Persona IQ Cohort: The study device is intended to relieve pain and restore function in patients with adequate quality and quantity of bone stock to support the prosthesis.
  The device is indicated for use in patients undergoing a cemented TKA that are normally indicated for at least a 30 mm sized tibial stem extension and/or normally indicated for at least a 58mm sized tibial stem.
  To qualify to receive the CTE/CSE with CHIRP System, the patient must be a candidate for commercially available Persona IQ Personalized Knee System implanted in accordance with product labeling.
  Interventions: Device: Persona IQ

INTERVENTIONS:
Device: Persona IQ — Persona IQ is a system comprised of the following subsystems:
  1. RTM utilizing mymobility® patient application and care team dashboard,
  2. PPK System with
  3. CTE Extension Implant and Instrumentation,
     1. Surgical Base Station System,
     2. Home Base Station System,
     3. Canary CDMP,
     4. Canary CMGP software module, and
  4. The ZBEdgeTM Connected Artificial Intelligence data platform.
  The system combines physical components, electronics, software, and user interfaces to collect, store, analyze, transmit, and display patient data for use by both physicians and patients.

SUMMARY:
A prospective multicenter longitudinal cohort study of Zimmer Biomet (ZB) Persona IQ The Smart Knee which consists of the Persona Personalized Knee (PPK) System with mymobility® platform that is attempting to develop correlative measures to assist surgeons in understanding and managing risk in their patient populations. Specifically comparing kinematic metrics captured via Remote Therapeutic Monitoring (RTM) utilizing the CANARY canturio te (CTE) and canturio se (CSE) sensors in combination with the mymobility® App.

The purpose of this study is to evaluate safety, functional performance, and effectiveness of the implant.

Primary Objective:

Assess Persona IQ kinematic metrics captured via the CTE/CSE sensor to assist surgeons in understanding and managing recovery through post-operative gait metrics.

Secondary Objective:

Evaluate the value of Remote Therapeutic Monitoring (RTM) and healthcare utilization.

Exploratory Objective:

Exploratory analyses will be performed using these data to direct future product feature development, data algorithm products, and research. This includes but is not limited to participants implanted utilizing ROSA® Robotics and other ZBEdge technologies.

DETAILED DESCRIPTION:
The Canary Tibial Extension (CTE)/canturio Smart Extension (CSE) with Canary Health Implanted Reporting Processor (CHIRP) System are intended to provide objective kinematic data from the implanted medical device during a patient's total knee arthroplasty (TKA) post-surgical care. The kinematic data are an adjunct to other physiological parameter measurement tools applied or utilized by the physician during the course of patient monitoring and treatment post-surgery.

The device is indicated for use in patients undergoing a cemented TKA procedure that are normally indicated for at least a 30 mm sized tibial stem extension and/or normally indicated for at least a 58mm sized tibial stem extension. The objective kinematic data generated by the CTE/CSE with CHIRP System are not intended to support clinical decision-making and have not been shown to provide any clinical benefit. The CTE/CSE with CHIRP System is compatible with Zimmer Persona® Personalized Knee System

The CTE/CSE with CHIRP System uses external OR and Home Base Station units to query the CTE/CSE implant (which has an internal radio and antenna) and upload the data collected by the CTE/CSE implant to the Canary Cloud data management platform (CDMP). Information from the implant is processed by the system's Canary Medical Gait Parameter (CMGP) software, located in the Cloud, into clinically relevant metrics.

Follow-up Procedures:

Follow-up evaluations will be conducted at 1 month (± 14 days), 3 months (± 30 days), and 1 year (± 90 days) after surgery. The 1-year visit will be optional. At every follow-up visit, pain and function of the study knee will be evaluated, and subject's quality of life will be assessed.

RTM assessments will be collected pre-operatively and post-operatively through the mymobility® care plan pathway as defined within the application for each specified assessment. The interval window will open and close automatically within the software for each specified target and captured clinically up-to 1-year post-operatively and indefinitely if the patient continues to utilize the mymobility App. Data will also be captured via the CTE/CSE sensors at variable intervals post-operatively and transmit data indefinitely if the home base station is connected and has power.

Data collected through mymobility® will include, but is not limited to the following:

* KOOS, JR
* EQ-5D-5L
* FJS-12
* Pain & Opioid Tracking

Data collected passively through CTE/CSE Sensors will include, but is not limited to the following:

* Walking Speed
* Cadence
* Stride Length
* Functional Knee ROM
* Tibial ROM
* Step Count
* Distance Traveled In-Person clinical assessments will be collected at 1-month, 3-months, and 1-year (optional).

Clinical Data Collection: The Sponsor will collect all data within multiple databases (e.g. including but not limited to: EDC, mymobility®, HealthKit, Google Fit, PIQ, ROSA). The management of all study data received by the Sponsor will be the responsibility of the Sponsor or its designee. The use or disclosure of all protected health information will comply with all relevant data privacy and data security laws and requirements. All information will be treated with strict adherence to professional standards of confidentiality and will be held by the Sponsor under adequate security and restricted accessibility.

Sample Size Calculation:

The study objective is to assess the seven kinematic metrics (step count, functional knee ROM, tibial ROM, distance walked, walking speed, cadence and stride length) to be captured via the CTE/CSE sensor in combination with the mymobility® platform and develop correlative insights to assist surgeons in understanding and managing recovery in their patient populations through post-operative gait metrics. All the clinical outcomes and device safety data to be collected will be summarized by the applicable univariate statistics and analyzed by the appropriate statistical models. In general, the logistic regressions for the categorical data point, especially binary data for rare events such as revision, hospital readmission etc., tend to require relatively large sample sizes to have enough power to perform conclusive analyses. According to Bujang et al. [5], 100 + 50i patients are needed to effectively use logistics regression in predicting outcomes, where i refers to the number of independent variables in the final model. It is expected between 15 and 20 independent variables will be available for the model. Assuming 18 independent variables, the sample size needs to be n = 1,000.

General Statistical Methods:

Data collected in this study will be summarized descriptively. Categorical data (such as biological sex, complications, satisfaction status, etc.) will be summarized using counts and percentages over the time periods of interest. Continuous data (such as age, ROM, etc.) will be summarized by using means, medians, standard deviation, minimum, maximum, and 95% CI over the time periods of interest.

Appropriate linear regression and generalized linear regression models including logistic regression, cox regression, mixed model for repeated measurements will be applied for the primary, secondary and exploratory endpoints analysis per the data type and analysis goals. Subgroup analysis on a variety of subsets of the collected data will also be performed. The applied statistical models will be used to evaluate and quantify the relationship among the differences in the episode of care data, patient pre-op physical condition and medical history, gait parameters, range of motion, patient satisfaction, nine most common post TKR complication incident rates, PROs, etc. Implant survival will be evaluated using Kaplan-Meier product limit estimate and raw survival rates. In addition to inference models, the predictive models will also be built to predict the patient satisfaction and PROs using patient baseline status and early PIQ data.

Data Analysis:

Primary Endpoints: The primary endpoints based on the clinical outcomes of the Canary Smart Tibial Stem when used in conjunction with the Persona IQ and mymobility® Platform for primary total knee arthroplasty will be analyzed by the appropriate linear and generalized linear regression models per the data type prospectively. The descriptive statistics will be provided as needed to individually describe the data points. The incidence of the most common post TKR medical complications will be analyzed by binary logistic regression model and time to event model such as cox regression. The relationship between pre-op, episode of care and post-operative gait recoveries will be evaluated by both binary logistic regression model and mixed model. The correlation between continuous 14 to 30-days Persona IQ data and 90-days post-operative sagittal ROM data will be evaluated by Pearson correlation, Intraclass Correlation Coefficient (ICC) with and without patient key baseline features adjusted. The relationship between categorical 14 to 30-days Persona IQ data and 90-days post-operative sagittal ROM data will be evaluated by either ANOVA or ANCOVA model per the analysis goal. The ordinary logistic regression will be applied to build predicting model for patient satisfaction at 42 and 90-days.

Secondary Endpoints: The evaluation of value related to the use of Remote Therapeutic Monitoring and healthcare utilization in the form of non-standard of care surgeon office visits, post-operative physical therapy, emergency department visits, and hospital readmissions associated with the index procedure will be evaluated using descriptive statistics as described in Section 16.2 along with appropriate statistical models.

Exploratory Endpoints: Implant survival and safety will be analyzed by Kaplan-Meier product limit estimate and raw survival rates with 95% confidence interval. Patient functional performance, clinical benefit measurements and healthcare utilization with index procedure will be analyzed for the whole cohort and for varied subgroups stratified by important surgical or clinical or patient physical features via both appropriate statistical models and descriptive statistics. The continuous clinical outcome differences between the subjects utilizing ROSA and conventional implantation will be evaluated by ANCOVA model with baseline function score, patient key baseline features and visit time adjusted. Other statistical methods will be utilized as appropriate to address the exploratory hypotheses.

ELIGIBILITY:
Inclusion Criteria

* Patient must be 18 years of age or older.
* Patient qualifies for primary unilateral, staged bilateral or simultaneous bilateral total knee arthroplasty.
* Independent of study participation, patient is a candidate for commercially available Persona IQ Personalized Knee System implanted in accordance with product labeling.
* Patient has access to appropriate technology to ensure full functionality for the home base station used as a part of their study procedure.
* Patient has access to the mymobility platform via eligible smart device.
* Patient must be willing and able to complete the protocol required follow-up.
* Patient is willing and able to provide written Informed Consent and Authorization by signing and dating the IRB approved Informed Consent and Authorization form.
* Patient is able to read and understand the language used in the mymobility app for their region.

Exclusion Criteria

* Patient is a current alcohol or drug abuser.
* Patient is known to be pregnant, breastfeeding, or considered a member of a protected class (e.g., prisoner, mentally incompetent, etc.).
* Patient has a psychiatric illness or cognitive deficit that will not allow proper informed consent and participation in follow-up program.
* Patient is currently participating in any other surgical intervention study which would compromise the results of this study, as determined by the Investigator.
* Patient has previous history of infection in the affected joint and/or other local/systemic infection that may affect the prosthetic joint.
* Patient has Neuropathic Arthropathy.
* Patient has osteoporosis, or any loss of musculature or neuromuscular disease that compromises the affected limb, as determined by the Investigator.
* Patient has gout, or a history of gout in the affected knee.
* Patient is undergoing procedures or treatments using ionizing radiation at or in the proximity of the CTE/CSE.
* Off-label use or not according to the approved instructions for use (IFU) of study devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The device is indicated for use in patients undergoing a cemented TKA procedure that are normally indicated for at least a 30 mm sized tibial stem extension and/or normally indicated for at least a 58mm sized tibial stem extension.
  In order to qualify to receive the CTE/CSE with CHIRP system, the patient must meet the following requirements in addition to any requirements for TKA surgery as determined by the patient's surgeon:
  1. The Patient's anatomy must be capable of accepting the Zimmer Biomet Persona Tibial Baseplate with CTE/CSE construct sizing. This assessment will be conducted pre-operatively by the surgeon using a CTE/CSE X-ray Template available through your Zimmer Biomet Representative.
  2. The patient must have access to a computer with a USB connection to set up their Home Base Station or have access to a compatible smartphone to set up their Home Base Station (Bluetooth).
  3. The Patient must have wireless internet in their domicile.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
mymobility platform data compared to most common AEs. | 1 year
  Assess the differences in episode of care, data compiled, collected, and delivered in the mymobility platform to correlate the incidence of nine most common post TKR medical complications. Nine most common post TKR medical complications: wound complication, thromboembolic disease, neural deficit, vascular injury, medial collateral ligament injury, instability, malalignment, stiffness, deep periprosthetic joint infection.
mymobility platform data compared to CTE/CSE data. | 1 year
  Comparison of mymobility platform data gait analysis to CTE data gait analysis.
Identify 14 to 30-days Persona IQ data points which correlate with 90-days post op full, arthrokinematic sagittal ROM data. | 90 days
  Functional ROM during a qualified gait cycle. Calculated from tibia ROM. Mean sagittal plane functional ROM when walking. Difference between maximum and minimum knee joint flexion.
mymobility platform data combined with CTE/CSE data compared to patient satisfaction at various intervals post op. | 1 year
  Assess the ability of post-op data compiled, collected, and delivered in the mymobility application (from, among other sources, the patient's smartphone sensors and Persona IQ implant data) collected during PODs 0-90 to predict which subjects will have a "very satisfied" or "satisfied" score on the Patient Satisfaction at 42 and 90-days.
  Potential Sources of Data: Smartphone Agnostic (iPhone or Android).Captures Google Fit steps from Android phone (and Fitbit, if data is imported to Google Fit app in Android application) as well as HealthKit Mobility Metrics from qualified iOS devices (steps, stairs, gait speed, asymmetry, etc.).
  Smartphone, Smartwatch, and PIQ activity dashboards displayed in surgeon/care team dashboard (Web or Mobile) and in patient app experience (Web or Mobile).
  Modular functionality allows care team to select content and management feature customization.

SECONDARY OUTCOMES:
Full patient clinical, mymobility platform data combined with CTE as it pertains to bearing variants at various intervals post op. | 1 year
  Utilize the unique patient clinical data that is available with the mymobility application to correlate early post-operative outcomes of ZB bearing component variants ultracongruent (UC), cruciate retaining (CR), medial congruent (MC), posterior stabilized (PS) & constrained posterior stabilized (CPS) to pre-operative and post-operative activity profiles, surgical techniques, patient attributes, and other routine outcomes data collected.
Full patient clinical, mymobility platform data combined with CTE data analysis for future product feature development. | 1 year
  To provide a real-world data set on the Persona IQ / mymobility cohort, including physiologic monitoring data, that enables ongoing exploratory data analysis and retrospective cohort study that will inform future product feature development, data algorithm products, and research. An example of such analysis that would support surgeons to make patient-specific recommendations is: pre-operative patient phenotype risk profiling combined with an "early stiffness detection" that could lead toward a triage care pathway progressions.

OTHER OUTCOMES:
Implant survival measured in years. | 1 year
Implant safety measured in frequency of adverse events. | 1 year
Functional performance measured through patient reported outcome measures total scores via Knee Injury and Osteoarthritis Outcome Score - Short Form (KOOS, JR). | 1 year
Functional performance measured through patient reported outcome measures total scores via Lower Extremity Functional Scale (LEFS). | 1 year
Functional performance measured through patient reported outcome measures total scores via Forgotten Joint Score (FJS-12). | 1 year
Functional performance measured through patient reported outcome measures total scores via EuroQol-5 Dimensions-5 Levels - Health-Related Quality of Life Survey (EQ-5D-5L). | 1 year
Rate of healthcare utilization in the form of non-standard of care surgeon office visits, post-operative physical therapy, emergency department visits and hospital readmissions associated with the index procedure. | 1 year
Number of subjects implanted utilizing ROSA compared to the number of subjects that underwent conventional implantation. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Erin Osborn, Study Director — Zimmer Biomet
Locations (4):
- United States (4):
  - Jeffrey Yergler, LLC/South Bend Orthopaedics, Granger, Indiana
  - Washington University, St Louis, Missouri
  - OrthoCarolina Research Institute, Charlotte, North Carolina
  - Rothman Institute, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided